CLINICAL TRIAL: NCT00836147
Title: A Single-centre, Double Blind, Randomised, Exploratory Study to Explore the Efficacy and Safety of Juvista 250ng/100µL/Linear cm When Administered Following Excision of Ear Lobe Keloids.
Brief Title: Exploratory Study of the Efficacy and Safety of Juvista 250ng When Administered Following Excision of Ear Lobe Keloids
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Renovo (Industry)
Responsible Party: Amanda Hilton Senior Clinical Research Manager, Renovo Ltd
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: RN1001-0107
Record Dates: First submitted 2009-02-03; First posted 2009-02-04 (Estimated); Last update posted 2010-09-28 (Estimated); Status verified 2010-09

CONDITIONS: Keloid
MeSH Terms: conditions — Keloid | interventions — TGFB3 protein, human

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Placebo Comparator): 250 ng dose
  Interventions: Drug: Avotermin (Juvista)
- 2 (Active Comparator): 250 ng dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Avotermin (Juvista) — 20 patients undergoing surgical revision of bilateral ear lobe keloids. Injecting intradermally 250ng/100µL/linear cm of the wound margin to one ear lobe and placebo into the other wound margin immediately after surgery and then 24hrs after wound closure.
  Arms: 1
Drug: Placebo — 20 patients undergoing surgical revision of bilateral ear lobe keloids. Injecting intradermally 250ng/100µL/linear cm of the wound margin to one ear lobe and placebo into the other wound margin immediately after surgery and then 24hrs after wound closure.
  Arms: 2

SUMMARY:
This trial will explore the efficacy and safety of 250ng Juvista per Linear cm, administered by intradermal injection following the excision of ear lobe keloids. Keloids commonly occur after ear piercing and are usually bilateral.One ear lobe will be treated with Juvist and one with placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-85 years who have given written informed consent.
* Subjects with bilateral ear lobe keloid scars of comparable size and suitable for surgical excision which will result in a single wound on each ear lobe no greater than 2cm long and restricted to the skin, fat and fibrous tissue of the ear lobe.
* Subjects with, in the opinion of the investigator, clinically acceptable results for the laboratory tests specified in the trial protocol (see Protocol Section 6.3.2). All laboratory tests must be performed within 28 days of the first trial dose administration.
* Female subjects of child bearing potential who are using a highly effective method(s) of contraception and agree to do so from at least the screening visit until one month after administration of the final study dose. For the purposes of the protocol, highly effective method(s) of contraception will be defined as consistently and correctly used implants, injectables, combined oral contraceptives, sexual abstinence or a vasectomised partner.

Exclusion Criteria:

* Subjects who have had ear lobe keloids treated with irradiation, cryosurgery, corticosteroids, or other pharmacological agents in the three months prior to the first trial dose administration.
* Subjects with a history of a bleeding disorder.
* Subjects who on direct questioning and/or physical examination have past or present evidence of eczema or psoriasis local to the site of administration, uncontrolled diabetes (fasting plasma glucose concentration consistently at or above 7.0mmol 1-1 (126 mg dl-1), severely immunocompromised patients and/or malignant skin tumours e.g. melanomas, squamous or basal cell carcinomas.
* Subjects with a skin disorder, not related to the keloid disease, that is chronic or currently active and which the Investigator considers will adversely affect the healing of the acute wounds or involves the areas to be examined in this trial.
* Subjects with a history of malignancy in the last 5 years.
* Subjects with a history of hypersensitivity to any of the drugs or dressings used in this trial.
* Subjects who are taking, or have taken any investigational product or participated in a clinical trial in the three months prior to first trial dose administration.
* Subjects undergoing investigations or changes in management for an existing medical condition.
* Subjects who, in the opinion of the Investigator, are unlikely to complete the trial for whatever reason.
* Female subjects who are pregnant or lactating.
* Subjects with a creatinine clearance (CLcr) of 80ml/min or less. Creatinine clearance will be determined from the serum creatinine level at pre-study screening using the following formula.

CLcr = 140 - age (years) x Weight (kg) 72 x serum creatinine mg/dL [ x 0.85 for females]

* Subjects who are not able to undergo MRI scanning due to their medical history or physical condition.
* Subjects who have previously received treatment with Juvista (Avotermin).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2009-02; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Keloid recurrance | 12 months

SECONDARY OUTCOMES:
Frequency of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: V. Leroy Young, MD, Principal Investigator — Body Aesthetic Plastic Surgery and Skincare Center, St Louis, Missori, United States
Locations (1):
- Body Aesthetic Plastic Surgery and Skincare Center, St Louis, Missouri, United States